CLINICAL TRIAL: NCT01020825
Title: A Prospective Study for the Assessment of the Long-term Safety and Efficacy of Cx401 in Patients Taking Part in the FATT-1 Trial
Brief Title: Long-term Safety and Efficacy of Adipose-derived Stem Cells to Treat Complex Perianal Fistulas in Patients Participating in the FATT-1 Randomized Controlled Trial
Acronym: LTE
Status: Completed | Type: Observational
Sponsor: Tigenix S.A.U. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: CX401-0303; EudraCT: 2008-003140-10 (Other: EMEA)
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Complex Perianal Fistula
Keywords: Complex perianal fistula; Adipose-derived adult stem cells; Fibrin glue
MeSH Terms: interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ASCs: Patients randomized to experimental treatment (ASC transplantation) in the FATT-1 randomized controlled trial [ClinicalTrials.gov identifier: NTC00475410]
  Interventions: Drug: ASCs
- Fibrin glue: Patients randomized to the control treatment (application of fibrin glue) in the FATT-1 randomized controlled trial [ClinicalTrials.gov identifier: NTC00475410]
  Interventions: Drug: Fibrin glue
- ASCs + Fibrin Glue: Patients randomized to the control treatment (application of fibrin glue) + intralesional injection of ASCs in the FATT-1 randomized controlled trial [ClinicalTrials.gov identifier: NTC00475410]
  Interventions: Drug: ASCs

INTERVENTIONS:
Drug: ASCs — Intralesional injection of adult-stem-cells at a dose of 20 and 40 million.
  Other Names: Cx401 (company code); Ontaril®
  Groups: ASCs
Drug: Fibrin glue — After curettage, the fistulous tract was sealed with fibrin glue.
  Groups: Fibrin glue
Drug: ASCs — Intralesional injection of adult-stem-cells at a dose of 20 and 40 million in combination with fibrin glue.
  Other Names: Cx401 (company code); Ontaril®
  Groups: ASCs + Fibrin Glue

SUMMARY:
The purpose of this extension is to investigate and confirm the long-term (6 months) safety and efficacy of the preceding FATT-1 trial [ClinicalTrials.gov identifier: NTC00475410], which studied patients with perianal fistula treated having received adipose-derived adult stem cell (ASC)and/or fibrin glue.

DETAILED DESCRIPTION:
Complex perianal fistulas are a source of great distress for suffers. Treatment options are limited and surgery is often associated with incontinence and recurrence.

The biological properties of stem cells derived from adult tissues make them candidates for the treatment of pathologies requiring tissue regeneration or in diseases where the healing process is altered.

This study aims to evaluate the safety and efficacy of patients having participated within a preceding multicenter, placebo-controlled, phase 3 study [ClinicalTrials.gov identifier: NTC00475410]. The present extension aims to collect safety and efficacy data for up to 12 month from initial administration.

Fistula closure is defined as absence of suppuration through the external orifice with complete re-epithelization of the external orifice and absence of collections >2cm directly related to the fistula tract treated, as measured by MRI.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 dose of the treatment assigned in the FATT-1 trial
* Informed consent

Exclusion Criteria:

* Other experimental drugs other than Cx401 during the follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that received at least one treatment dose in study Cx401/FATT1
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of adverse events (clinical or laboratory) attributed to the study therapy in the preceding FATT-1 randomized trial (CX401 or fibrin glue) | 6 months (since last visit in FATT-1 trial)

SECONDARY OUTCOMES:
Closure of the fistula (defined as suppuration through the external opening of the fistula spontaneously and on pressure, complete re-epithelization of the external opening in the clinical evaluation and absence of collections >2 cm in MRI) | 6 months (since last visit of FATT-1 trial)

CONTACTS AND LOCATIONS:
Overall Officials: Damián García-Olmo, MD, Principal Investigator — General Surgery Department, Hospital Universitario La Paz
Locations (15):
- Spain (15):
  - Hospital Mutua de Terrasa, Terrassa, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Doctor Josep Trueta, Girona
  - Hospital Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clínica Universitaria Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora de Valme, Seville
  - Hospital Universitari Joan XXIII, Tarragona
  - Hospital General Univeritario de Valencia, Valencia
  - Hospital Clínico Universitario "Lozano Blesa", Zaragoza

REFERENCES:
- [Background] Garcia-Olmo D, Garcia-Arranz M, Garcia LG, Cuellar ES, Blanco IF, Prianes LA, Montes JA, Pinto FL, Marcos DH, Garcia-Sancho L. Autologous stem cell transplantation for treatment of rectovaginal fistula in perianal Crohn's disease: a new cell-based therapy. Int J Colorectal Dis. 2003 Sep;18(5):451-4. doi: 10.1007/s00384-003-0490-3. Epub 2003 May 20. PMID 12756590
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D, Pascual I, Peiro C, Rodriguez-Montes JA. A phase I clinical trial of the treatment of Crohn's fistula by adipose mesenchymal stem cell transplantation. Dis Colon Rectum. 2005 Jul;48(7):1416-23. doi: 10.1007/s10350-005-0052-6. PMID 15933795
- [Background] Garcia-Olmo D, Herreros D, Pascual M, Pascual I, De-La-Quintana P, Trebol J, Garcia-Arranz M. Treatment of enterocutaneous fistula in Crohn's Disease with adipose-derived stem cells: a comparison of protocols with and without cell expansion. Int J Colorectal Dis. 2009 Jan;24(1):27-30. doi: 10.1007/s00384-008-0559-0. Epub 2008 Aug 12. PMID 18696086
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D. Expanded adipose-derived stem cells for the treatment of complex perianal fistula including Crohn's disease. Expert Opin Biol Ther. 2008 Sep;8(9):1417-23. doi: 10.1517/14712598.8.9.1417. PMID 18694359
- [Derived] Herreros MD, Garcia-Arranz M, Guadalajara H, De-La-Quintana P, Garcia-Olmo D; FATT Collaborative Group. Autologous expanded adipose-derived stem cells for the treatment of complex cryptoglandular perianal fistulas: a phase III randomized clinical trial (FATT 1: fistula Advanced Therapy Trial 1) and long-term evaluation. Dis Colon Rectum. 2012 Jul;55(7):762-72. doi: 10.1097/DCR.0b013e318255364a. PMID 22706128